CLINICAL TRIAL: NCT04236713
Title: Evaluation of Food Additive Contributions to Obesity - Feasibility Study 3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Natalia McInnes, Associate Professor, McMaster University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7992
Record Dates: First submitted 2020-01-04; First posted 2020-01-22 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention 1 (Experimental)
  Interventions: Other: Dietary intervention 1
- Dietary intervention 2 (Experimental)
  Interventions: Other: Dietary intervention 2

INTERVENTIONS:
Other: Dietary intervention 1 — Limiting dietary exposure to ethylenediaminetetraacetic acid, erythorbate, propionate and related food additives; limiting eating out to a maximum of 2 days per week.
  Arms: Dietary intervention 1
Other: Dietary intervention 2 — Limiting dietary exposure to nitrites, sulfites and related food additives; limiting eating out to a maximum of 2 days per week; limiting drinking wine to a maximum of 2 days per week.
  Arms: Dietary intervention 2

SUMMARY:
The effects of food additives on body weight in humans are largely unknown. This is a feasibility study in 10 obese adults who will be followed for 5 months. Eligible participants will be non-randomly assigned to 2 groups and will be taught how to limit the exposure to the studied food additives in their diet. Primary outcomes in this study are recruitment rate, retention rate and adherence to the proposed dietary intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI >/=30 kg/m2
* willingness and ability to follow the proposed dietary interventions
* informed consent

Exclusion Criteria:

* previous or planned bariatric surgery in the next 1 year
* current or planned participation in any structured weight-loss programs in the next 6 months
* current or recent (within the last 6 months) use of weight-loss-inducing drugs or systemic steroids
* excessive alcohol consumption
* bipolar disorder or attention deficit hyperactivity disorder
* current use of anti-depressant or anti-psychotic medications
* eating disorder or any other active disorder that may lead to significant weight changes
* pregnancy or planned pregnancy in the next 1 year
* uncontrolled diabetes mellitus or diabetes requiring treatment with >2 oral diabetes medications or with insulin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 0 months
  Average number of participants recruited per month
Retention rate in arm 1 | 5 months
  Percent of enrolled participants who complete the study
Retention rate in arm 2 | 5 months
  Percent of enrolled participants who complete the study
Adherence to the dietary intervention in arm 1 | 2 to 5 months
  Proportion of meals/beverages free of the studied food additives on 3 unannounced 24-hour dietary recalls
Adherence to the dietary intervention in arm 2 | 2 to 5 months
  Proportion of meals/beverages free of the studied food additives on 3 unannounced 24-hour dietary recalls

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No